CLINICAL TRIAL: NCT04776447
Title: A Phase II Trial of Atezolizumab Plus Induction Chemotherapy (CT) Plus Chemo-radiotherapy and Atezolizumab Maintenance Therapy in Non-resectable Stage IIIA-IIIB Non-small Cell Lung Cancer (NSCLC) Patients
Brief Title: Atezolizumab Plus Induction Chemotherapy Plus CT-radiotherapy. (APOLO)
Acronym: APOLO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 20/08_APOLO; 2020-004459-33 (EudraCT Number)
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Lung Diseases; Carcinoma, Non-Small-Cell Lung; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Respiratory Tract Neoplasms; Carcinoma Bronchiogenic Stage III; Thoracic Neoplasms
Keywords: Chemo-radiotherapy; Immunotherapy; Atezolizumab; Carboplatin; Paclitaxel; Induction chemotherapy; Maintenance treatment; ctDNA levels; Antineoplastic Agents; Induction chemo-immunotherapy; Non-resectable non-small cell lung cancer
MeSH Terms: conditions — Lung Diseases; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Carcinoma, Bronchogenic; Thoracic Neoplasms | interventions — Carboplatin; Paclitaxel; atezolizumab

STUDY DESIGN:
Intervention Model Description: Design: Open-label, non-randomized, phase II multi-centre controlled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Atezolizumab plus induction chemotherapy plus CT-radiotherapy (Experimental): Induction Treatment:
  Atezolizumab: 1200mg, IV infusion Carboplatin: AUC5, IV infusion Paclitaxel: 200 mg/m2 The treatment will start within 1-5 days from enrollment. The treatment will be 3 cycles administered at 21-day intervals.
  Concurrent Chemotherapy (CT)-Radiotherapy Treatment:
  Chemotherapy and radiotherapy treatment will be at the discretion of the principal investigator of each site. It is recommended to use as concurrent chemotherapy treatment a platinum based doublet.
  After the 3rd cycle of the induction treatment, concurrent treatment will start, 1st concurrent cycle will be administered from day 1 of cycle 3 of induction treatment.
  Concurrent chest radiotherapy will be administered starting at day 1 of cycle 1 of concurrent chemo-radiotherapy.
  Maintenance with Atezolizumab:
  Atezolizumab: 1200mg, IV infusion After the 3rd cycle of the concurrent treatment, Atezolizumab maintenance treatment will start from day 1 of cycle 6 and will be administered for 12 months.
  Interventions: Drug: Carboplatin; Drug: Placlitaxel; Drug: Atezolizumab

INTERVENTIONS:
Drug: Carboplatin — Structure: The cis-diamino (cyclobutane-1, 1 dicarboxylate) plating. Stability: 24 hours at ambient temperature in 5% glucose, glucosamine or physiologic saline. It is recommended not to dilute with chlorinated solutions for this could affect the carboplatin.
  Route of administration: Intravenous infusion.
  Guidelines of Carboplatin administration: According to the standard of each center.
  Other Name: ATC code: L01XA02
  Other Names: Carboplatinum
Drug: Placlitaxel — Structure: A diterpene whose composition is: 5b, 20-epoxy-1, 2a, 4,7b, 10b, 13a-hexahidroxytax-11-en 9 one 4,10-diacetate 2-benzoate 13-ester with (2R,3S)- N-benzoyl-3-phenylisoserine.
  Stability: Concentrations of 0.3-1.2 mg/ml in 5% dextrose or normal saline have demonstrated chemical and physical stability for more than 27 hours at ambient temperature (25ºC approximately). The intact vial must be stored between 15º and 25ºC.
  Guidelines of Paclitaxel administration: Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  Other Names: Taxol
Drug: Atezolizumab — Atezolizumab is a humanized immunoglobulin (IgG1) monoclonal antibody that is produced in Chinese hamster ovary (CHO) cells. Atezolizumab targets programmed death-ligand 1 (PD-L1) on tumor-infiltrating immune cells (ICs) or tumor cells (TCs) and prevents interaction with the programmed death-1 (PD-1) receptor and B7.1 (CD80), both of which function as inhibitory receptors expressed on T cells and other immune cells.
  Patients will receive 1200 mg of atezolizumab administered by IV infusion every 21 days (+/- 3 days) in a monitored setting where there is immediate access to trained personnel and adequate equipment/medicine to manage potentially serious reactions.
  Other Names: Tecentriq

SUMMARY:
Open-label, non-randomized, phase II multi-centre controlled clinical trial.

51 non-resectable stage IIIA-IIIB non-small cell lung cancer patients will be enrolled in this trial to evaluate the efficacy of the treatment (Atezolizumab + Induction chemotherapy (CT) + CT-Radiotherapy) in terms of the Progression Free Survival at 12 months

DETAILED DESCRIPTION:
This is an open-label, non-randomized, phase II multi-centre controlled clinical trial.The total sample size is 51 patients. The population to be included are non-resectable stage IIIA-IIIB non-small cell lung cancer patients.

Patients randomised will receive induction treatment (Atezolizumab 1200mg+ Carboplatin AUC5+Paclitaxel 200 mg/m2 for 3 cycles) and concurrent chemotherapy (CT) -radiotherapy treatment for 3 cycles. At the end of concurrent treatment Atezolizumab 1200mg maintenance treatment will start and will be administered for 12 months (16 cycles).

The primary objective is to assess the efficacy of the treatment (Atezolizumab + Induction chemotherapy (CT) + CT-Radiotherapy) in terms of the Progression Free Survival (PFS) at 12 months according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.

PFS are defined as the time from inclusion until objective tumor progression or death.

Patient accrual is expected to be completed within 2 years, treatment is planned to extend during 1.5 years and the patients will be followed up for 2 years. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years old and ≤ 75 years.
* ECOG Scale (Eastern Cooperative Oncology Group) of performance status of 0 or 1.
* Histologically or cytologically confirmed, non-resectable Stage IIIA-IIIB NSCLC according to the 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology.
* PET-CT (Positron Emission Tomography -Computed tomography) and brain computed tomography or Magnetic resonance imaging (MRI) at baseline to confirm the absence of distant disease.
* Mediastinal involvement could be considered without histological confirmation when no margin can be distinguished in the lymph node mass.
* No prior treatment with anti-neoplastic drugs or thoracic radiotherapy for Stage IIIA-IIIB NSCLC.
* Patients who have received prior neo-adjuvant, adjuvant chemotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from enrollment since the last chemotherapy.
* Presence of at least one measurable disease by CT-SCAN, as defined by RECIST v1.1.
* Adequate hematologic and organ function defined by the following laboratory results obtained within 14 days prior to enrollment:
* Neutrophils ≥ 1500 cells/μL without granulocyte colony-stimulating factor support.
* Lymphocyte count ≥ 500/μL.
* Platelet count ≥ 100,000/μL without transfusion.
* Haemoglobin ≥ 10.0 g/dL. Patients may be transfused to meet this criterion.
* INR or aPTT ≤ 1.5 × upper limit of normal (ULN). This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
* AST, ALT, and alkaline phosphatase ≤ 2.5 × ULN, with the following exceptions:
* Serum bilirubin ≤ 1.5 × ULN. Patients with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled.
* Serum creatinine ≤ 1.5 × ULN or creatinine clearance of ≥60ml/min (based on the Cockcroft Gault formula).
* All patients are notified of the investigational nature of this study and signed a written informed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention.
* Adequate lung function: Forced Expiratory Volumen in 1 second (FEV1) >50% of normal volume and Diffusion Capacity of the Lungs for Carbon Monoxide (DLCO) >40% of normal value.
* No more than 35% of the total volume of the two lungs should receive more than 20 Gy (V20) or no more than 7cm maximum diameter.
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate (< 1% per year) when used consistently and correctly, and to continue its use for 6 months after the last dose of trial treatment. Such methods include: combined (oestrogen and progesterone containing) hormonal contraception, progestogen-only hormonal contraception associated with inhibition of ovulation together with another additional barrier method always containing a spermicide, intrauterine device (IUD): intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner (on the understanding that this is the only one partner during the whole study duration), and sexual abstinence.
* For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception that results in a low failure rate [< 1% per year] when used consistently and correctly, and to continue its use for 6 months after the last dose of trial treatment. Male patients should not donate sperm during this study and for at least 6 months after the last dose of trial treatment.
* Oral contraception should always be combined with an additional contraceptive method because of a potential interaction with the study drugs. The same rules are valid for male patients involved in this clinical study if they have a partner of childbirth potential. Male patients must always use a condom.
* Women who are not postmenopausal (≥ 12 months of non-therapy-induced amenorrhea) or surgically sterile must have a negative serum pregnancy test result within 8 days prior to initiation of study drug.

Exclusion Criteria:

* Patients with known sensitizing mutation or an amplification in the epidermal growth factor receptor (EGFR) gene, ALK fusion oncogene.
* Known STK-11 ligand alterations, MDM2 amplifications or ROS1 translocations.
* Weight loss >10% within the previous 3 months.
* Malignant pleural effusion or pericardial effusion: both will be considered as suggestive of metastatic disease. Also excluded those with negative cytology but being exudates.
* Patients with non-visible by thoracic X-Ray pleural effusion or too small to be safely punctioned could be included.
* Malignancies other than NSCLC within 3 years prior to enrollment, with the exception of those with a negligible risk of metastasis or death (e.g., expected 3-year OS > 90%) treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous-cell skin cancer, localized prostate cancer treated with radiotherapy or surgically with curative intent, ductal carcinoma in situ treated surgically with curative intent).
* Women who are pregnant, lactating, or intending to become pregnant during the study.
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the Atezolizumab formulation.
* History of autoimmune disease.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
* Positive test for human immunodeficiency viruses (HIV). All patients will be tested for HIV prior to inclusion into the study; patients who test positive for HIV will be excluded from the clinical study.
* Patients with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.
* Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible only if they are negative for HBV DNA (vaccinated patients are excluded).
* Patients positive for hepatitis C virus (HCV) antibody are eligible only if PCR is negative for HCV RNA.
* Active tuberculosis.
* Symptomatic neuropathy (sensory) grade > 1 according to the NCI Common Toxicity Criteria for Adverse Events v5.0
* Severe infections within 4 weeks prior to be included in the study, including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
* Received therapeutic oral or IV antibiotics within 2 weeks prior to be included in the study.
* Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction, or cerebrovascular accident within 3 months prior to inclusion, unstable arrhythmias, or unstable angina.
* Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
* Patients with a superior vena cava syndrome.
* Major surgical procedure other than for diagnosis within 28 days prior to inclusion or anticipation of need for a major surgical procedure during the course of the study.
* Prior allogeneic bone marrow transplantation or solid organ transplant.
* Administration of a live, attenuated vaccine within 4 weeks before inclusion or anticipation that such a live attenuated vaccine will be required during the study.
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.
* Patients with illnesses or conditions that interfere with their capacity to understand follow and/or comply with study procedures.
* Treatment with any other investigational agent with therapeutic intent within 28 days prior to initiation of study treatment.
* Treatment with systemic immunosuppressive medications (including but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of the treatment in terms of the Progression Free Survival (PFS) at 12 months | From the date of the end of treatment until 12 months
  To assess the efficacy of the treatment (Atezolizumab + Induction chemotherapy (CT) + CT-Radiotherapy) in terms of the Progression Free Survival (PFS) at 12 months according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1.PFS is defined as the time from inclusion until objective tumor progression or death.

SECONDARY OUTCOMES:
To evaluate the Overall Response Rate (ORR) of the treatment | From the date of randomization to the date of last follow up, assessed up to 36 months
  To evaluate the ORR of the treatment as measured by investigator-assessed overall response rate (ORR) according to RECIST v1.1.
To evaluate the Overall survival (OS) rate | From the date of the end of treatment until 12 and 24 months
  To evaluate the Overall survival (OS) rate at 12 and 24 months of the treatment.
To evaluate the sites of first failure | From the date of the end of treatment until the date of last follow up, assessed up to 36 months
  To evaluate the sites of first relapse or progression
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 30 days after the final administration of the drug
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — Fundación GECP President
Locations (22):
- Spain (22):
  - Hospital General Universitario de Elche, Elche, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Insular de Gran canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Parc Taulí, Barcelona
  - Hospital de Basurto, Bilbao
  - ICO Girona, Hospital Josep Trueta, Girona
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Santa María Nai, Ourense
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Clínico de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org